CLINICAL TRIAL: NCT02243384
Title: A Randomized Controlled Trial of Laparoscopic Hepatectomy and Radiofrequency Ablation in the Treatment of Early Hepatocellular Carcinoma
Brief Title: Laparoscopic Hepatectomy and Radiofrequency Ablation in the Treatment of Early Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChenJian (Other)
Responsible Party: Sponsor-Investigator, ChenJian, Associate Professor of Hepatobiliary Surgery Institute; Chief Physician; Administrator of laparoscopic department, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: chenjian-01
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Early Hepatocellular Carcinoma; Laparoscopic Hepatectomy; Radiofrequency Ablation; Micrometastases
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Micrometastasis | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and researchers do not understand the test grouping, but the research designer arranges and controls all trials.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Hepatectomy (Experimental): Laparoscopic Hepatectomy
  Interventions: Procedure: Laparoscopic Hepatectomy
- Radiofrequency Ablation (Active Comparator): Radiofrequency Ablation
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Laparoscopic Hepatectomy — A total of 110 patients with early HCC with nodular diameters of less than 3 cm and up to three nodules were randomly divided into LH (n=55) and RFA groups (n=55). Outcomes were carefully monitored and evaluated during the 3-year follow-up period
  Arms: Laparoscopic Hepatectomy
Procedure: Radiofrequency Ablation — A total of 110 patients with early HCC with nodular diameters of less than 3 cm and up to three nodules were randomly divided into LH (n=55) and RFA groups (n=55). Outcomes were carefully monitored and evaluated during the 3-year follow-up period
  Arms: Radiofrequency Ablation

SUMMARY:
The purpose of this research is to compare short-term and long-term efficacy of laparoscopic hepatectomy and radiofrequency ablation in the Treatment of early hepatocellular carcinoma, and provide the evidence for the choice of surgical method from the pathology and cytology.

DETAILED DESCRIPTION:
Background:The aim of this study was to compare the efficacy of laparoscopic hepatectomy(LH) with radiofrequency ablation (RFA) in the treatment of early hepatocellular carcinoma (HCC).

Methods:A total of 110 patients with early HCC with nodular diameters of less than 3 cm and up to three nodules were randomly divided into LH (n=55) and RFA groups (n=55). Outcomes were carefully monitored and evaluated during the 3-year follow-up period.

Results:

operation time, intraoperative blood loss, rate of blood transfusion, complications and mortality, postoperative liver function, resection margin, number of micrometastases ,long-term curative effect and survival time were collected and analysed.

groups t-test ，univariate/multivariate analysis, logistic regression analysis, mixed linear regression, Cox survival analysis ，Kaplan-Meier survival analysis，Log-rank survival curves were used.

ELIGIBILITY:
Inclusion Criteria:

* Any gender,18 to 70 years old;
* Preoperative diagnosis of primary liver clear;
* No active hepatitis and decompensated cirrhosis;
* Maximum diameter ≤3cm single nodules or three nodules in diameter and no more than 3cm,did not infringe the portal vein,hepatic vein and inferior vena cava invasion,lymph node or extrahepatic turn;
* No tumor rupture or bleeding;
* Child-Pugh class A or B grade,ICG-R15 <14%;
* No coagulation disorders,platelet count > 50 × 109 / L and prolonged prothrombin time < 5 seconds;
* Not be including related surgery,radiofrequency ablation (RFA),TACE treatment,no certainty anticancer chemotherapy treatment;supreme absolute contraindications abdominal surgery;
* Patients generally available,heart and lung function can tolerate surgery, abdominal surgery supreme absolute contraindications;
* Voluntarily participate in the study,informed consent.

Exclusion Criteria:

* Age < 18 years or > 70,pregnant and lactating women;
* Primary liver cancer diagnosis is not clear
* Liver function assessment:Child-PughC level,liver function reserve situation :ICGR-15> 14%
* Tumor rupture has occurred,or has the line before surgery,radiofrequency ablation (RFA),TACE or chemotherapy cancer treatment;
* Tips liver imaging with multiple ( > 3 ) lesion,or tumor diameter> 3 cm, clear portal vein,hepatic vein,inferior vena cava tumor thrombus trunk;
* Preoperative liver metastasis;
* Preoperative evaluation of cardiopulmonary dysfunction patients who can not tolerate surgery;
* Intraoperative exploration has occurred disseminated tumor and / or lymph node metastasis;
* Exploratory surgery found that non-hepatic primary tumors,such as colorectal metastases,hilar cell carcinoma;
* Severe upper abdominal adhesions;
* Postoperative pathological examination of the bile duct cell or mixed cell carcinoma and pathologically confirmed positive margin;
* Foreign,Hong Kong,Macao,Taiwan and other regions,estimated postoperative difficult to track,followed up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Survival rate | 5 years
  follow-up after the surgery every 2 months, to understand relapse, death, statistics 1 year, 2-year and 3-year survival, disease-free survival, recurrence rate.

SECONDARY OUTCOMES:
postoperative complications | Duration hospitalization(an expected average of 7 days)
  hepatic failure,hemorrhage,biliary leakage,ascites,intra-abdominal infection,pleural effusion,pulmonary infection,cardiac insufficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Chen, Study Chair — Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- JianChen, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Result] Amarapurkar D, Han KH, Chan HL, Ueno Y; Asia-Pacific Working Party on Prevention of Hepatocellular Carcinoma. Application of surveillance programs for hepatocellular carcinoma in the Asia-Pacific Region. J Gastroenterol Hepatol. 2009 Jun;24(6):955-61. doi: 10.1111/j.1440-1746.2009.05805.x. Epub 2009 Mar 11. PMID 19383082
- [Result] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Result] Jarnagin W, Chapman WC, Curley S, D'Angelica M, Rosen C, Dixon E, Nagorney D; American Hepato-Pancreato-Biliary Association; Society of Surgical Oncology; Society for Surgery of the Alimentary Tract. Surgical treatment of hepatocellular carcinoma: expert consensus statement. HPB (Oxford). 2010 Jun;12(5):302-10. doi: 10.1111/j.1477-2574.2010.00182.x. PMID 20590903
- [Result] Zimmerman MA, Ghobrial RM, Tong MJ, Hiatt JR, Cameron AM, Hong J, Busuttil RW. Recurrence of hepatocellular carcinoma following liver transplantation: a review of preoperative and postoperative prognostic indicators. Arch Surg. 2008 Feb;143(2):182-8; discussion 188. doi: 10.1001/archsurg.2007.39. PMID 18283144
- [Result] Reich H, McGlynn F, DeCaprio J, Budin R. Laparoscopic excision of benign liver lesions. Obstet Gynecol. 1991 Nov;78(5 Pt 2):956-8. PMID 1833688
- [Result] Kobayashi T. Long-term Survival Analysis of Pure Laparoscopic Versus Open Hepatectomy for Hepatocellular Carcinoma in Patients With Cirrhosis: A Single-center Experience. Ann Surg. 2015 Jul;262(1):e20. doi: 10.1097/SLA.0000000000000443. No abstract available. PMID 24368662
- [Result] Zhou YM, Shao WY, Zhao YF, Xu DH, Li B. Meta-analysis of laparoscopic versus open resection for hepatocellular carcinoma. Dig Dis Sci. 2011 Jul;56(7):1937-43. doi: 10.1007/s10620-011-1572-7. Epub 2011 Jan 23. PMID 21259071
- [Result] Nguyen KT, Marsh JW, Tsung A, Steel JJ, Gamblin TC, Geller DA. Comparative benefits of laparoscopic vs open hepatic resection: a critical appraisal. Arch Surg. 2011 Mar;146(3):348-56. doi: 10.1001/archsurg.2010.248. Epub 2010 Nov 15. PMID 21079109
- [Result] Cherqui D, Husson E, Hammoud R, Malassagne B, Stephan F, Bensaid S, Rotman N, Fagniez PL. Laparoscopic liver resections: a feasibility study in 30 patients. Ann Surg. 2000 Dec;232(6):753-62. doi: 10.1097/00000658-200012000-00004. PMID 11088070
- [Result] Otsuka Y, Tsuchiya M, Maeda T, Katagiri T, Isii J, Tamura A, Yamazaki K, Kubota Y, Suzuki T, Suzuki T, Kagami S, Kaneko H. Laparoscopic hepatectomy for liver tumors: proposals for standardization. J Hepatobiliary Pancreat Surg. 2009;16(6):720-5. doi: 10.1007/s00534-009-0139-x. Epub 2009 Aug 4. PMID 19652902
- [Result] Ishizawa T, Gumbs AA, Kokudo N, Gayet B. Laparoscopic segmentectomy of the liver: from segment I to VIII. Ann Surg. 2012 Dec;256(6):959-64. doi: 10.1097/SLA.0b013e31825ffed3. PMID 22968066
- [Result] Dagher I, Belli G, Fantini C, Laurent A, Tayar C, Lainas P, Tranchart H, Franco D, Cherqui D. Laparoscopic hepatectomy for hepatocellular carcinoma: a European experience. J Am Coll Surg. 2010 Jul;211(1):16-23. doi: 10.1016/j.jamcollsurg.2010.03.012. Epub 2010 May 26. PMID 20610244
- [Result] Livraghi T. Radiofrequency ablation of hepatocellular carcinoma. Surg Oncol Clin N Am. 2011 Apr;20(2):281-99, viii. doi: 10.1016/j.soc.2010.11.010. PMID 21377584
- [Result] Lau WY, Lai EC. The current role of radiofrequency ablation in the management of hepatocellular carcinoma: a systematic review. Ann Surg. 2009 Jan;249(1):20-5. doi: 10.1097/SLA.0b013e31818eec29. PMID 19106671
- [Result] Mulier S, Ni Y, Jamart J, Ruers T, Marchal G, Michel L. Local recurrence after hepatic radiofrequency coagulation: multivariate meta-analysis and review of contributing factors. Ann Surg. 2005 Aug;242(2):158-71. doi: 10.1097/01.sla.0000171032.99149.fe. PMID 16041205
- [Result] Feng K, Yan J, Li X, Xia F, Ma K, Wang S, Bie P, Dong J. A randomized controlled trial of radiofrequency ablation and surgical resection in the treatment of small hepatocellular carcinoma. J Hepatol. 2012 Oct;57(4):794-802. doi: 10.1016/j.jhep.2012.05.007. Epub 2012 May 23. PMID 22634125
- [Result] Buell JF, Cherqui D, Geller DA, O'Rourke N, Iannitti D, Dagher I, Koffron AJ, Thomas M, Gayet B, Han HS, Wakabayashi G, Belli G, Kaneko H, Ker CG, Scatton O, Laurent A, Abdalla EK, Chaudhury P, Dutson E, Gamblin C, D'Angelica M, Nagorney D, Testa G, Labow D, Manas D, Poon RT, Nelson H, Martin R, Clary B, Pinson WC, Martinie J, Vauthey JN, Goldstein R, Roayaie S, Barlet D, Espat J, Abecassis M, Rees M, Fong Y, McMasters KM, Broelsch C, Busuttil R, Belghiti J, Strasberg S, Chari RS; World Consensus Conference on Laparoscopic Surgery. The international position on laparoscopic liver surgery: The Louisville Statement, 2008. Ann Surg. 2009 Nov;250(5):825-30. doi: 10.1097/sla.0b013e3181b3b2d8. PMID 19916210
- [Result] Yin Z, Fan X, Ye H, Yin D, Wang J. Short- and long-term outcomes after laparoscopic and open hepatectomy for hepatocellular carcinoma: a global systematic review and meta-analysis. Ann Surg Oncol. 2013 Apr;20(4):1203-15. doi: 10.1245/s10434-012-2705-8. Epub 2012 Oct 26. PMID 23099728
- [Result] Katz SC, Shia J, Liau KH, Gonen M, Ruo L, Jarnagin WR, Fong Y, D'Angelica MI, Blumgart LH, Dematteo RP. Operative blood loss independently predicts recurrence and survival after resection of hepatocellular carcinoma. Ann Surg. 2009 Apr;249(4):617-23. doi: 10.1097/SLA.0b013e31819ed22f. PMID 19300227
- [Result] Minami Y, Kudo M. Radiofrequency ablation of hepatocellular carcinoma: Current status. World J Radiol. 2010 Nov 28;2(11):417-24. doi: 10.4329/wjr.v2.i11.417. PMID 21179308
- [Result] Shi M, Guo RP, Lin XJ, Zhang YQ, Chen MS, Zhang CQ, Lau WY, Li JQ. Partial hepatectomy with wide versus narrow resection margin for solitary hepatocellular carcinoma: a prospective randomized trial. Ann Surg. 2007 Jan;245(1):36-43. doi: 10.1097/01.sla.0000231758.07868.71. PMID 17197963
- [Result] Curley SA. Radiofrequency ablation leads to excellent local tumor control and durable longterm survival in specific subsets of early stage HCC patients confirming to the Milan criteria. Ann Surg. 2010 Dec;252(6):913-4. doi: 10.1097/SLA.0b013e3182034862. No abstract available. PMID 21107101
- [Result] Huang J, Yan L, Cheng Z, Wu H, Du L, Wang J, Xu Y, Zeng Y. A randomized trial comparing radiofrequency ablation and surgical resection for HCC conforming to the Milan criteria. Ann Surg. 2010 Dec;252(6):903-12. doi: 10.1097/SLA.0b013e3181efc656. PMID 21107100
- [Derived] Song J, Cao L, Ma K, Li J, Wang X, Chen J, Zheng S. Laparoscopic liver resection versus radiofrequency ablation for small hepatocellular carcinoma: randomized clinical trial. Br J Surg. 2024 Apr 3;111(4):znae099. doi: 10.1093/bjs/znae099. PMID 38650579